CLINICAL TRIAL: NCT04013464
Title: Changes of Sleep EEG Power and Melatonin Rhythm in Major Depressive Disoder: a Self-controlled, 8 Weeks Study of Treatment With Escitalopram Compared With Healthy Subjects
Brief Title: Effects of Escitalopram on the Sleep EEG Power in Patients With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Sixth Hospital (Other)
Collaborators: National Institute on Drug Dependence, China (Other)
Responsible Party: Principal Investigator, Xueqin Wang, Associate professor, M.D., Peking University Sixth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-4-2113
Record Dates: First submitted 2019-06-26; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Intervention Model Description: Major depressive disorder compared to health control
Masking Description: changed into escitalopram in open treatment and compared to health control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MDD and Health Control (Experimental): MDD in open label
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10-20mg/d
  Other Names: no other intervention

SUMMARY:
The main objective was to compare the differences of PSG parameters and plasma melatonin levels before and after treatment with escitalopram for 8 weeks. Polysomnography (PSG) was detected over a night and blood samples were collected at 4 h intervals for 24 h from 13 male healthy controls and 13 male MDD patients before and after treatment with escitalopram for 8 weeks. The outcome measures included the levels of plasma melatonin, PSG parameters (include sleep architecture and power analysis) and scales.

DETAILED DESCRIPTION:
1. Design and participants: The patients with MDD were screened from the hospital, age- and gender-matched healthy controls were recruited by advertising from the community who signed written informed consent before participation.
2. Assessments: The 17-item Hamilton Depression Rating Scale (HRSD-17) , Montgomery-Asberg Depression Rating Scale (MADRS), the Clinical Global Impression-Severity scale (CGI-S), and 14-item Hamilton anxiety scale (HAMA) were assessed at baseline and after 8 weeks' treatment with escitalopram for patients with MDD. As for healthy volunteer, these measures were evaluated only once. In addition, all participants were assessed Pittsburgh Sleep Quality Index (PSQI) and Insomnia Severity Index (ISI).
3. Treatment: Each patient was provided with escitalopram.
4. Collection of peripheral blood samples: Test the levels of plasma melatonin at 4 h intervals for 24 h from all participants.
5. Sleep and EEG recordings: The PSG of participants was evaluated for one night at baseline (all participants) and 8 weeks treatment (MDD).
6. Analysis the PSG architecture and power ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of MDD;
2. Hamilton Rating Scale for Depression 17-items (HRSD-17) total scores ≥ 22;
3. Male patients aged between 18 and 45 years

Exclusion Criteria:

1. Significant suicide risk by HRSD suicide scores > 2;
2. Accompanied with psychiatric symptoms;
3. Treated with MECT within 6 months.

Ages: 22 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy of MDD in the treatment of escitalopram | 8 weeks
  The 17-item Hamilton Depression Rating Scale (HRSD-17) was defined a prior as the primary outcome measure .
Sleep ratio of EEG power changes in MDD after 8 weeks treatment by escitalopram | 8 weeks
  polysomnography (PSG) was detected over a night and power analysis was done.
The levels changes of plasma melatonin after 8 weeks treatment by escitalopram | 8 weeks
  Test the levels of plasma melatonin at 7 time points during 24 h in MDD.

CONTACTS AND LOCATIONS:
Overall Officials: Su-Xia Li, Doctor, Principal Investigator — National Institute on Drug Dependence, China

IPD SHARING:
Plan to Share IPD: No